CLINICAL TRIAL: NCT02756104
Title: T Cell Phenotypes in ALS, Influence of Vitamin D
Brief Title: T Cell Phenotypes in Amyotropic Lateral Sclerosis (ALS), Influence of Vitamin D
Acronym: VITALS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Collaborators: ARSLA (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 9632
Record Dates: First submitted 2016-04-18; First posted 2016-04-29 (Estimated); Last update posted 2020-05-29 (Actual); Status verified 2020-05

CONDITIONS: ALS
MeSH Terms: interventions — Dietary Supplements; Vitamin D

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Volunteers (Other): Healthy People on each collecting blood for phenotyping Tcells
  Interventions: Other: phenotyping Tcells
- Patients with ALS (Other): Patients with ALS deficient or not in Vitamin D on each collecting blood for phenotyping Tcells.
  The patients who are deficient in Vitamin D will have supplementation in vitamin D
  Interventions: Other: phenotyping Tcells; Other: Supplementation in vitamin D

INTERVENTIONS:
Other: phenotyping Tcells — Collecting blood for analyses of the T cells phenotypes
Other: Supplementation in vitamin D — Supplementation in vitamin D for the patients who are deficient on vitamin D
  Arms: Patients with ALS

SUMMARY:
ALS is a devastative disorder characterized by motor neuron degeneration. Median survival is 3 years after onset, but may vary from a few months to more than 30 years. Various factors have been suspected to play a role in such a variation, but recently, it has been described that regulatory T-lymphocytes (T regs) may mediate ALS progression and survival. Vitamin D is an hormone know to regulated T reg function in vivo and in vitro. It have recently demonstrated that vitamin D (VD) levels correlated with ALS prognosis. The investigator want to go further in the study of the immune processes that could modulate prognosis in ALS. This could allow proposing VD as a potential treatment of ALS in a future trial. More largely, this could reinforce arguments in favor of an immune intervention to attenuate the severity of this devastating disorder.

DETAILED DESCRIPTION:
ALS is a devastative disorder characterized by motor neuron degeneration. Median survival is 3 years after onset, but may vary from a few months to more than 30 years. Various factors have been suspected to play a role in such a variation, but recently, it has been described that regulatory T-lymphocytes (T regs) may mediate ALS progression and survival. Vitamin D is an hormone know to regulated T reg function in vivo and in vitro. It have recently demonstrated that vitamin D (VD) levels correlated with ALS prognosis and patients with a severe VD deficiency had a 6 time more rapid evolution than those with normal VD levels. The investigator want to go further in the study of the immune processes that could modulate prognosis in ALS. We propose 1- to study T cell phenotypes (Treg, CD4 (cluster of differentiation 4) -Th1, -Th17, -Th2, CD8 (cluster of differentiation 8)and NK) in ALS vs controls ; 2- In VD-deficient patients, to analyze the influence of a vitamin D supplementation on T cell phenotypes ; 3- to study the relationships between T cell phenotypes and ALS prognostic factors. The project will include 70 ALS patients and 27 controls in this prospective study. VD-deficient patients will be supplemented, according to national recommendations for 6 months, and the evolution of T cell phenotypes will be followed over 1 year. We hope to demonstrate first that T cell phenotypes in ALS are consistent with a pro inflammatory profile, compared to controls, secondly that VD treatment modulates T cell phenotypes towards a non-inflammatory one and, thirdly, that inflammatory T cell phenotypes correlate with a worse prognosis of the disease. This could allow proposing VD as a potential treatment of ALS in a future trial. More largely, this could reinforce arguments in favor of an immune intervention to attenuate the severity of this devastating disorder.

ELIGIBILITY:
For the patients :

Inclusion Criteria:

* Man or woman with sporadic ALS and a possible, probable or definite diagnosis regarding the revised Escorial criteria (Forbes et al., 2001). Patients are followed quarterly according to national recommendations. At the end of the follow up period (1 year for each patient), all patients remaining in the " possible " group of diagnosis will be excluded.
* Disease onset (date of onset of muscle weakness) < 18 months at the time of inclusion.
* Age: 30 to 80 years-old, inclusive.
* Patient treated by riluzole at a steady dosage since at least 3 months.
* Patient accepting to give informed consent

Exclusion criteria will be :

* A previous treatment with VD in the preceding 2 years, whatever the dose used.
* Patient with an already known autoimmune disorder
* Patient with severe ALS involvement suggesting that survival over the 1 year follow up is highly unlikely (ex : tetraplegia, use of non-invasive ventilation for more than 10 hrs/day, ALSFRS-R (ALS Functional Rating Scale) score < à 20).
* Pregnant or breast-feeding woman.
* Patient without social security insurance

For the Controls:

Controls will be spouses of our ALS patients. Such a group has the advantage of similar life style conditions, and frequently similar geographical origin. Controls and ALS patients will match for age and gender. Controls will also fulfill the following inclusion and exclusion criteria

Inclusion criteria

•Subject accepting to give informed consent

Exclusion criteria

* Subject with an already known neurodegenerative disorder
* Subject with an already known autoimmune disorder
* Subject who received a treatment with VD in the preceding 2 years, whatever the dose used.
* Pregnant or breastfeeding woman
* Subject without social security insurance

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2016-06-07 (Actual); Primary Completion 2018-09-10 (Actual); Study Completion 2020-05-25 (Actual)

PRIMARY OUTCOMES:
Study of T-cell phenotypes in ALS patients and controls | 6 months
  Analyses of the expression of T cells phenotypes between volunteers and patients with ALS

SECONDARY OUTCOMES:
Influence of vitamin D treatment on T cell phenotypes | 6 months
  Study the relation between vitamin D blood level and the lymphocytes phenotypes between patient with initial ALS and volunteers
Relationships between expression of T cell phenotypes and ALS criteria | 6 months
  Study of the relation between the lymphocytes phenotypes expression and prognostic factors of the ALS
Relationships between vitamin D blood level and pronostic factors of the ALS | 6 months
  Study of the relation between vitamin D blood level and prognostic factors of the ALS

CONTACTS AND LOCATIONS:
Overall Officials: William CAMU, MD/PhD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- University Hospital of Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Yes
The investigator communicate the global results on demand